CLINICAL TRIAL: NCT02547636
Title: Prospective Clinical Evaluation of the FilmArray® NGDS Warrior Panel
Status: Completed | Type: Observational
Sponsor: BioFire Diagnostics, LLC (Industry)
Collaborators: BioFire Defense LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: DX-SDY-020450
Record Dates: First submitted 2015-09-10; First posted 2015-09-11 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Evaluation of Test Panel
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residual specimens may be stored for use as negative clinical matrix in contrived testing studies.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects/specimens that meet the inclusion criteria: Subjects/specimens that meet the inclusion criteria
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — No intervention will be used in this study.

SUMMARY:
This study will evaluate the clinical specificity of the FilmArray NGDS Warrior Panel.

ELIGIBILITY:
Inclusion Criteria:

* Whole blood (prospectively collected via informed consent):
* Adult subject has a recorded or self-reported fever within the previous 24 hours
* Subject provides informed consent prior to enrollment and specimen collection
* Subject has not previously provided a whole blood specimen for this study

Whole blood (residual)

* Whole blood (in EDTA) submitted to laboratory for standard of care testing
* Specimen is not from an individual with a specimen previously enrolled in the study

Positive Blood Culture:

* Culture was detected as positive by an automated blood culture system
* Culture is not from a patient previously enrolled in the study

Negative Blood Culture:

* Culture not detected as positive by an automated blood culture system
* Culture is not from a patient previously enrolled in the study

Sputum:

* Specimen was accepted for testing by the respective site's microbiology laboratory
* Specimen is not from an individual that has a sputum already enrolled in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with fever will be prospectively enrolled, and whole blood will be collected. Additional residual specimens left-over from standard of care laboratory testing will also be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 1822 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Clinical specificity of the FilmArray NGDS Warrior Panel | 8 months

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Navy Medical Center San Diego/Naval Health Research Center, San Diego, California
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Washington University/Barnes Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Ohio State University Medical Center, Columbus, Ohio
  - Madigan Army Medical Center, Tacoma, Washington